CLINICAL TRIAL: NCT06410313
Title: First In Human Study to Assess Safety and Efficacy of the ChampioNIR™ Drug Eluting Peripheral Stent in the Treatment of Patients With Superficial Femoral Artery Disease and/or Proximal Popliteal Artery Disease
Acronym: CHAMPIONSHIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medinol Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChampioNIR DES-001
Record Dates: First submitted 2024-05-01; First posted 2024-05-13 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Superficial Femoral Artery Stenosis; Popliteal Artery Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- ChampioNIR™ Ridaforolimus Eluting Peripheral Stent System (Experimental): ChampioNIR™ Ridaforolimus Eluting Peripheral Stent System
  Interventions: Device: ChampioNIR Ridaforolimus Eluting Peripheral Stent System

INTERVENTIONS:
Device: ChampioNIR Ridaforolimus Eluting Peripheral Stent System — ChampioNIR implantation in Patients with Superficial Femoral Artery Disease and/or Proximal Popliteal Artery disease

SUMMARY:
This is a prospective, open label, multicenter, single arm, first in human clinical study.

Patients with infra-inguinal peripheral arterial disease appropriate for treatment with a femoro-popliteal stent will be enrolled. The patients will be treated with the ChampioNIR Stent System. All implanted patients will be followed up at 30 days and 6, 12, 24 and 36 months. The follow-up visits will include patency evaluation by duplex ultrasound

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and of age of legal consent.
2. Subject has lifestyle limiting claudication or rest pain (Rutherford-Becker scale 2-4) with a resting ankle-brachial index/toe-brachial index (ABI/TBI) <0.90/0.80.
3. A single superficial femoral artery lesion with >50% stenosis or total occlusion.
4. Stenotic lesion(s) or occluded length within the same vessel (one long or multiple serial lesions) ≤ 150 mm.
5. Reference vessel diameter (RVD) ≥ 3.0 mm and ≤ 5.0 mm by visual assessment.
6. Target lesion located with the distal point at least 3 cm above the knee joint, defined as the distal end of the femur at the knee joint, and proximal point at least 2 cm below the origin of the profunda femoris (deep femoral artery).
7. Patent infra-popliteal and popliteal artery, i.e., single vessel runoff or better with at least one of three vessels patent (<50% stenosis) to the ankle or foot.
8. The target lesion(s) can be successfully crossed with a guide wire and dilated.
9. The subject is eligible for standard surgical repair, if necessary.
10. Subjects are willing to comply with scheduled visits and tests and are able and willing to provide informed consent.

Exclusion Criteria:

1. Presence of thrombus in the treated vessel as visualized by angiography, prior to crossing the lesion.
2. Thrombolysis of the target vessel within 72 hours prior to the index procedure, where complete resolution of the thrombus was not achieved.
3. Poor aortoiliac or common femoral "inflow" (i.e. angiographically defined >50% stenosis of the iliac or common femoral artery) that would be deemed inadequate to support a femoro-popliteal bypass graft and was not successfully treated prior to treatment of the target lesion either within the same procedure or at least 30 days prior to the index procedure.
4. Presence of residual ≥30% stenosis after either PTA or stenting of the inflow lesion.
5. Presence of an ipsilateral arterial artificial graft.
6. Ipsilateral femoral aneurysm or aneurysm in the SFA or popliteal artery.
7. Lesions in contralateral SFA/PPA that require intervention during the index procedure, or within 30 days before or after the index procedure;
8. Required stent placement (in the target or any other lesion) via a retrograde approach.
9. Required stent placement (in the target or any other lesion) across or within 0.5 cm of the SFA / PFA bifurcation.
10. Procedures which are pre-determined to require stent-in-stent placement to obtain patency, such as in-stent restenosis.
11. Significant vessel tortuosity or other parameters prohibiting access to the lesion or 90° tortuosity which would prevent delivery of the stent device.
12. Required stent placement within 1 cm of a previously (in a former procedure) deployed stent.
13. Use of atherectomy or other atheroablative (e.g. cryoplasty) devices at the time of index procedure.
14. Restenotic lesion that had previously been treated by atherectomy, laser or cryoplasty within 3 months of the index procedure.
15. Subject has tissue loss, defined as Rutherford-Becker classification category 5 or 6.
16. Overlapping stents are not allowed.
17. Coronary intervention within 7 days prior to or planned within 30 days after the treatment of the target lesion.
18. Stroke within the previous 30 days of the index procedure.
19. Known allergies to any of the following: aspirin, P2Y12 inhibitors (clopidogrel bisulfate, prasugrel, OR ticagrelor), heparin OR bivalirudin, nitinol (nickel titanium), PDLG, PLC, PDL, limus drugs (ridaforolimus, zotarolimus, tacrolimus, sirolimus, everolimus, or similar drugs or any other analogue or derivative or similar compounds) or contrast agent, that cannot be medically managed.
20. Receiving dialysis or immunosuppressant therapy within the previous 30 days.
21. Known or suspected active systemic infection at the time of the procedure.
22. Known bleeding or hypercoagulability disorder or significant anemia (Hb<8.0) that cannot be corrected.
23. Platelet count <50,000/μL
24. International normalized ratio (INR) > 1.5
25. GFR <30 ml/min by Cockroft-Gault.
26. Subject has a co-morbid illness that may result in a life expectancy of less than 1 year.
27. Planned use of a drug coated balloon (DCB) during the index procedure.
28. Pregnant women or women of childbearing potential who do not have a negative serum or urine pregnancy test documented within 7 days prior to enrollment.
29. Subject is participating in any investigational study that has not yet reached its primary endpoint

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Primary patency of the target lesion | 6 months
  Primary patency of the target lesion defined as the absence of target lesion restenosis (defined by Duplex ultrasound (US) peak systolic velocity ratio (PSVR) ≥2.4).
Primary safety endpoint | 30 days
  Composite rate of freedom from all-cause death, target vessel revascularization or any amputation of the index limb through 30 days following stent implantation

SECONDARY OUTCOMES:
Primary patency | 30 days and 12 months
  Primary patency defined by Duplex US peak systolic velocity ratio (absence of restenosis which defined by Duplex US PSVR ≥2.4)
Acute device success | During the index procedure
  Acute device success, defined as achievement of a final residual diameter stenosis of <30% by Quantitative Angiography (QA), using the assigned treatment only
Acute procedural success | During the index procedure
  Acute procedural success, defined as device success with <30% residual stenosis immediately after stent placement or mean trans-stenotic pressure gradient <5 mmHg, and without the occurrence of death, amputation or repeat revascularization of the target lesion during the hospital stay
Acute technical success | During the index procedure
  Acute technical success, defined as the attainment of <30% residual stenosis by QA by any percutaneous method as determined by the angiographic core laboratory
Secondary Patency | 30 days 6, 12, 24 and 36 months
  Secondary Patency (absence of restenosis which is defined as Duplex US PSVR ≥ 2.4)
Change of Rutherford classification | 30 days 6, 12, 24 and 36 months
  Change of Rutherford classification from baseline
Change of resting ankle-brachial index (ABI) | 30 days 6, 12, 24 and 36 months
  Change of resting ankle-brachial index (ABI) from baseline
Change in walking impairment questionnaire | 30 days 6, 12, 24 and 36 months
  Change in walking impairment questionnaire from baseline
Combined rate of the following events: death at 30 days, target vessel revascularization (TVR), index limb amputation and increase in Rutherford-Becker Classification by ≥2 classes (as compared to post-procedural assessment) | 12 months
  Combined rate of the following events:death at 30 days, target vessel revascularization (TVR), index limb amputation and increase in Rutherford-Becker Classification by ≥2 classes (as compared to post-procedural assessment)
Stent fracture | 12 and 36 months
  Evidence of Stent fracture analyzed by a two-view X-ray evaluation
Freedom from all-cause death, index limb amputation above the ankle and Target Vessel Revascularization | 30 days
  Freedom from all-cause death, index limb amputation above the ankle and Target Vessel Revascularization
All-cause death | 30 days, 6, 12, 24 and 36 months
  All-cause death
Amputation (above the ankle)-Free Survival (AFS) | 30 days, 6, 12, 24 and 36 months
  Amputation (above the ankle)-Free Survival (AFS)
Target Vessel Revascularization (TVR) | 30 days, 6, 12, 24 and 36 months
  Target Vessel Revascularization (TVR)
Target Lesion Revascularization (TLR) | 30 days, 6, 12, 24 and 36 months
  Target Lesion Revascularization (TLR)
Rate of Re-intervention for treatment of thrombosis of the target vessel or embolization to its distal vasculature | 30 days, 6, 12, 24 and 36 months
  Rate of Re-intervention for treatment of thrombosis of the target vessel or embolization to its distal vasculature
Major Adverse Limb Events (MALE) | 30 days, 6, 12, 24 and 36 months
  Stent thrombosis, Clinically apparent distal embolization, Procedure-related arterial rupture, Acute limb ischemia, Target limb amputation, Procedure related bleeding event requiring transfusion

CONTACTS AND LOCATIONS:
Locations (7):
- United States (3):
  - Piedmont Healthcare, Inc., Atlanta, Georgia
  - Columbia University Medical Center/ NewYork Presbyterian Hospital or CUMC/NYPH, New York, New York
  - St Francis Hospital Heart Center, Roslyn, New York
- Australia (4):
  - The Alfred Hospital, Melbourne
  - Royal Perth Hospital, Perth
  - Royal North Shore Hospital, Sydney
  - Royal Prince Alfred Hospital, Sydney

IPD SHARING:
Plan to Share IPD: No